CLINICAL TRIAL: NCT01491087
Title: Safety of the DTacP-IPV//PRP~T Combined Vaccine (PENTAXIM®) Given as a Three-Dose Primary Vaccination at 2, 3, and 4 Months of Age in Infants in China
Brief Title: Safety of PENTAXIM® Given as a Three-Dose Primary Vaccination at 2, 3, and 4 Months of Age in Infants in China
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: E2I60; U1111-1117-7233 (Other: WHO)
Record Dates: First submitted 2011-12-09; First posted 2011-12-13 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Diphtheria; Tetanus; Pertussis; Polio
Keywords: Pentaxim®; Whole-cell Pertussis vaccine; Acellular Pertussis vaccine; Haemophilus influenzae type b polysaccharide; Inactivated Polio vaccine; Pentavac®
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Poliomyelitis | interventions — Pentavac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PENTAXIM® vaccine group (Experimental)
  Interventions: Biological: DTacP IPV//PRP~T combined vaccine: PENTAXIM®

INTERVENTIONS:
Biological: DTacP IPV//PRP~T combined vaccine: PENTAXIM® — 0.5 mL, Intramuscular
  Other Names: PENTAXIM®

SUMMARY:
The study will assess the safety of Pentaxim® vaccine as a three-dose primary vaccination at 2, 3, and 4 months of age in order to meet the regulatory requirements for the license renewal as for any other product registered in China, and to generate additional clinical data using the three-dose primary vaccination schedule in some other Chinese provinces.

Primary Objective

* To describe the safety after administration of PENTAXIM® at 2, 3, and 4 months of age in the study population.

DETAILED DESCRIPTION:
Each study participant will receive an injection of PENTAXIM® at 2, 3, and 4 months of age and will be monitored for safety through the entire study period.

The duration of each participant in the trial will be approximately 3 to 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged 2 months (60 to 74 days) inclusive on the day of the first study visit
* Informed consent form has been signed and dated by the parent(s) or other legally acceptable representative
* Subject and parent/legally acceptable representative are able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* Participation or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy since birth, or long-term systemic corticosteroids therapy (prednisone or equivalent for more than 2 consecutive weeks since birth)
* Known systemic hypersensitivity to any of the vaccine components, or history of a life threatening reaction to the vaccine used in the trial or to a vaccine containing any of the same substances
* Clinically significant illness, according to investigator judgment, at a stage that could interfere with trial conduct or completion
* Evolving encephalopathy
* Receipt of immune globulins, blood or blood-derived products since birth
* Previous vaccination against diphtheria, tetanus, pertussis, poliomyelitis diseases or Haemophilus influenzae type b infection
* Receipt of any other vaccine in the 14 days preceding the first trial vaccination or planned receipt of any vaccine in the 14 days following the first trial vaccination
* Acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (axillary temperature ≥37.1°C). A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided.
* Contraindications to vaccination according to PENTAXIM® summary of product characteristics (SPC) or leaflet
* In an emergency setting, or hospitalized involuntarily
* Identified as a natural or adopted child of the Investigator or employee with direct involvement in the proposed study.

Ages: 60 Days to 74 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 900 (Actual)
Dates: Start 2011-12; Primary Completion 2012-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Description of the Safety profile in terms of solicited injection site and systemic reaction, and serious adverse events after each vaccination with PENTAXIM® vaccine | Day 0 for up to 3 months post vaccination
  Solicited injection site: Tenderness, Redness, and Swelling. Solicited Systemic reaction: Fever (Temperature), Vomiting, Abnormal crying, Drowsiness, Loss of Appetite, and Irritability

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (3):
- China (3):
  - Guangzhou, Guangdong
  - Shanghai
  - Tianjin

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com